CLINICAL TRIAL: NCT07142616
Title: Dignity Care - Digitally Supported Person-centered Care Systems
Brief Title: Digitally Supported Person-centered Care Systems
Acronym: DignityCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/ 251632
Record Dates: First submitted 2024-06-17; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Multiple Chronic Conditions
Keywords: Patient-Centered Care; Prevention; Integrated care; Electronic Health Records; Randomized controlled trial; Patient summary; Treatment plan; Decision Making, Shared
MeSH Terms: conditions — Multiple Chronic Conditions | interventions — Secondary Care

STUDY DESIGN:
Intervention Model Description: Participants are block randomized to balance the three arms (Usual care, 3 sources, Summaries). The sizes of the blocks are set by a trial service office, and not known to those involved in the trial.
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessor of the primary outcome is a large language model, which assesses the answers provided by the participants without any information about group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 01 Usual care with clinical notes from one provider (Active Comparator): Access to all clinical notes available to the provider in the patient's case. The provider is General practice in two patient cases, and hospital in one patient case.
  Interventions: Other: 01 - Clinical notes from one provider
- 02 Clinical notes from several providers (Active Comparator): Access to all clinical notes across three providers: General practitioner, Social services and Specialist care.
  Interventions: Other: 02 - Access to notes from primary and secondary care
- 03 - DigiTeam - Summaries of and clinical notes from several providers (Experimental): Access to all clinical notes across three providers: General practitioner, Social services and Specialist care, like in arm 02. In addition, access to information management features, such as summaries of patient's priorities, and clinical summaries of key health problems, including links to source documents.
  Interventions: Other: 03 - Summaries of and clinical notes from several providers

INTERVENTIONS:
Other: 03 - Summaries of and clinical notes from several providers — Access to all clinical notes across three providers: General practitioner, Social services and Specialist care, like in arm 02. In addition, access to information management features, such as summaries of patient's priorities, and clinical summaries of key health problems, including links to source documents.
  Arms: 03 - DigiTeam - Summaries of and clinical notes from several providers
Other: 01 - Clinical notes from one provider — Access to all clinical notes available to the provider in the patient's case. The provider is General practice in two patient cases, and hospital in one patient case.
  Arms: 01 Usual care with clinical notes from one provider
Other: 02 - Access to notes from primary and secondary care — Access to all clinical notes across three providers: General practitioner, Social services and Specialist care.
  Arms: 02 Clinical notes from several providers

SUMMARY:
The case history of patients with complex and long-term needs is often stored in fragments across many different care providers, each with a separate electronic health record. Even when the notes are stored in the same organization, the large volume of information makes it difficult for practitioners to grasp the full overview of the patient's situation.

The DigiTeam tool, combines information management features to present notes from across the care pathway from the three main providers: General Practice, Health and Social care Services, and Secondary care. It also includes summaries of the patient's concerns, conditions, and treatment plan. It provides links to the source documents that are the basis for the summaries.

The overarching aim is to examine the effect of physicians' use of the DigiTeam for three patient cases derived from real-world pseudonymized notes, on the quality of the physcians' ensuing case summary and treatment plan. In the comparator arms, physicians use usual care tools, i.e. only one or three sources of notes and no information management features.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner OR
* Physician who has graduated within the last five years.

If the recruitment is difficult, medical students and other physicians may be included.

To recruit participants, the trial will be announced through known networks, social media, the researchers' network, and general announcements.

Exclusion Criteria:

* There is no exclusion criterium.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of patient summary and follow-up plan | Immediately after completing the the task for each patient
  The primary outcome is the quality of the patient summary and follow-up plan
  Participants are asked to create a summary as preparation for a care planning meeting with colleagues, using the information available in the digital tool to write 1) a Comprehensive summary of the patient's situation and 2. A care plan.
  Quality of summaries and care plans will be measured by Microsoft Copilot. An expert group of three clinicians will create gold-standard summaries. These will be converted into a list of clear, mutually exclusive items using standardized rules. Copilot will be prompted to identify whether each item is present in participant responses. The item list will be validated by comparing scoring consistency (Kappa statistics) between researchers and Copilot, aiming for ≥0.7 agreement with researchers and ≥0.9 between Copilot runs. Final scores will reflect the number of items included per response.

SECONDARY OUTCOMES:
Time spent completeing the patient case overviews and follow-up plans | Immediately after completing the the task for each patient
  Time from start of case to delivery of answer as measured by participant reported start and stop time.
System Usability Scale | Immediately after completing the the task for each patient
  The usability of the intervention to do the work needed for each patient will be measured with the System Usability Scale which contains ten items scored from one (strongly disagree) to five (strongly agree) that are transformed to a 0 to 100 scale and translated into a curved grading scale from A-F
Information support for solving tasks | Immediately after completing the the task for each patient
  To compare how the different interventions helped to solve the task described under primary outcome, the following questions will be asked:
  On a scale of 1 to 5 (1 Poor 2 Fair 3 Good 4 Very good 5 Excellent), how did the information you had access to support you to find information about
  * Current medical status?
  * Social or personal circumstances that contribute to the current status?
  * What is important to the patient?
  * What should be followed up further?
  * Who should be involved in the follow-up?
Experience with conducting the task | Immediately after completing the the task for each patient
  To compare the experience with the digital tool used to conduct the tasks, the following questions will be used:
  On a scale of 1 to 5 (1 Poor 2 Fair 3 Good 4 Very good 5 Excellent)
  * What do you think about the tool overall?
  * How good was the support in the tool to find the information you needed?
  * How useful was the training in using the tool?
  * How did the tool work compared to tools you use daily for similar tasks?
  * How would such a tool fit into your daily work?
  Would you recommend the tool to colleagues? (Yes Unsure No)

OTHER OUTCOMES:
Technical problems | Immediately after completing the the task for each patient
  To describe the experience with the digital solution used, the following question will be used Did you have any technical problems in completing this task? No, none at all Some, but it was minimal Yes, quite extensive.
Experience with the type of patients | Immediately after completing the the task for each patient
  To describe whether the participants had experiences with the types of patients, the following question will be asked:
  How often do you work with patients who have as complex and long-term needs as this patient? (Weekly, Monthly, Semi-annually or less frequently)
Time spent on various activities | Immediately after completing the the task for each patient
  To describe the time used on various activities in the digital tool, the following variables will be automatically recorded in the tool:
  * Time spent in each main area: The main areas are the main pages in the side menu, like information about the patient, the list of clinical notes and the medication list.
  * Inactivity >10 seconds: The time the participant reads/writes.
  * Number of unique clinical notes that are opened.
  * Number of free text searches conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Gro KR Berntsen, Prof, Principal Investigator — Norwegian Center for E-health Research
Locations (1):
- University hospital North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized questionnaire data
Supporting Information: Study Protocol, ICF
Time Frame: At publication of planned papers from the RCT
Access Criteria: Contact authors.